CLINICAL TRIAL: NCT01161342
Title: Nutritional Status Among Older Adults. Risk Factors and Consequences of Malnutrition
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Principal Investigator, Lisa Söderström, Med.lic., Uppsala University
Other Study IDs: LTV-1211142
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2011-05

CONDITIONS: Malnutrition
Keywords: Malnutrition; Aged; Aged 80 and over; Prevalence; Mortality
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to estimate the prevalence of malnutrition among older adults admitted to hospital and to analyse predictive factors for malnutrition. Further, the aim was to analyse the association between nutritional status and all-cause and cause-specific mortality.

The hypothesis is that malnourished patients have a higher mortality then well-nourished patients after three years.

DETAILED DESCRIPTION:
The baseline survey was a cross-sectional study of 1771 patients aged ≥65 years who were admitted to hospital. Nutritional status was assessed using the MNA instrument, and possible risk factors associated with malnutrition were recorded during the hospital stay. All-cause mortality was followed up after median 3.5 years s in a cohort study of 1767 participants. Cause-specific mortality was followed up after median 4.7 years in a cohort of 1767 participants. Previous dietary intake in middle-aged and older adults was recorded at basline in 725 participants, who had their nutritional status assessed with the MNA when admitted to hospital 10 years later.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years or older

Exclusion Criteria:

* unable to communicate and no relative could anwer the questions (n = 356)
* receiving palliative care (n = 44)
* impossible to measure height or weight (n = 22)
* miscellanious (n = 71)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The included sample comprised 1771 patients 65 years and older, consecutively admitted during fifteen months to two internal medicine wards (n = 706), two surgical wards (n = 681), and one orthopaedic ward (n = 384) at the Central hospital in Västerås, Sweden.
Sampling Method: Probability Sample
Enrollment: 1771 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Nutritional status according to the screening instrument Mini Nutritional Assessment (MNA) | 30 minutes
  [The 18 questions in the MNA instrument are weighted, and the threshold values of the instrument categorize patients into three nutritional status groups: well-nourished (MNA score 24-30), at risk of malnutrition (MNA score 17-23.5), or malnourished (MNA score <17).
All-cause mortality | All-cause mortality was analyzed after median 3.5 years.
  Survival was calculated from the date of the MNA screening to the date of death.
Cause-specific mortality | Cause-specific mortality was analyzed after median 4.7 years.
  Survival was calculated from the date of the MNA screening to the date of cause-specific death.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bergkvist, Professor, Principal Investigator — The Center for Clinical research, the County Council of Vestmanland/Uppsala University, Sweden